CLINICAL TRIAL: NCT04093687
Title: Towards Painless Colonoscopy: a Dedicated Training to Decrease the Rate of Painful Colonoscopy - a Randomized Controlled Trial
Brief Title: Towards Painless Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Marek Bugajski, Principal Investigator, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MSCI
Record Dates: First submitted 2019-09-15; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Screening Colonoscopy; Pain During Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention will consist of one training session, focusing on technical and non-technical aspects identified in the study Phase I (according to the evaluation questionnaire). The training will be conducted by a team consisting of (i) supervisors (researchers) and (ii) teachers experienced in the previous trial (Train-Colonoscopy-Leaders course - TCL; this methodology has already been evaluated (citation)). There will be 7 trainees per session: 1 under-, 4 average and 2 overperformers.
  The training session will be divided into two parts: theoretical and practical. During the first, theoretical part of the training, the body of research on the phenomenon of colonoscopy pain will be presented. The second, practical part of the training, will consist of a one-day session of 7 colonoscopies.
  Each average and underperforming endoscopist who underwent training in the randomized phase will receive a written, customized feedback on his/her performance during the training session.
  Interventions: Other: Endoscopist's training
- Control Arm (No Intervention): The endoscopists in the control arm will not be informed about participation in the study and will receive only tailored feedback on adjusted painful colonoscopy rate (practice as usual). They will receive a reminder, that dedicated report on painful colonoscopy rate is provided in the Polish Colonoscopy Screening Program database and they will be monitored for endpoints through Polish Colonoscopy Screening Program database.

INTERVENTIONS:
Other: Endoscopist's training — The training session will be divided into two parts: theoretical and practical. Trainees will be blinded to the criterion of being chosen due to their performance status.
  During the first, theoretical part, the body of research on the phenomenon of colonoscopy pain will be presented. Aspects on how to deliver a painless colonoscopy (patient characteristics, insertion technique, endoscope characteristics, non-technical skills, additional manoeuvres) will be discussed. This part will be based on the findings from Phase I.
  The second, practical part of the training, will consist of a one-day session of 7 colonoscopies. Participants will be matched with each other. Each participant, will perform one colonoscopy with an oversight of a matched partner, then in turn oversee the colonoscopy of another participant. The rest of the participants will observe a live transmission of each colonoscopy in a separate room, with a commentary from study coordinator.
  Arms: Intervention Arm

SUMMARY:
One of the major barriers to CRC screening participation is a negative perception of colonoscopy as a painful and unpleasant procedure. Previously, by monitoring patient-reported outcomes as one of the colonoscopy quality performance measures, the investigators identified the endoscopist as the single, most important risk factor for painful colonoscopy. Therefore, the investigators propose a randomized controlled trial to analyse the effectiveness of directed training on the endoscopists painful colonoscopy rate.

The study will be conducted in two phases: endoscopist categorization and design of training (I) and randomized controlled trial evaluating training effectiveness (II).

Phase I will include endoscopists from Polish Colonoscopy Screening Programme (PCSP) willing to participate. Volunteers will be divided into underperformers, average performers and overperformers, based on their painful colonoscopy rate (obtained from PCSP database records) and will be invited to take part in the initial workshop focused on pain reduction during colonoscopy (conducted in a similar fashion to Train Colonoscopy Leaders (TCL) workshop, aiming at ADR improvement).

On the basis of the differences in performance between over- and underperformers, categories of importance, target scores and a questionnaire for the assessment of factors for improvement will be developed.

In Phase II, endoscopists from PCSP screening centres previously categorized as underperformers and average performers will be randomized in 1:1 ratio either to control (no intervention) or intervention arm.

The subjects in the control arm will not be trained or informed about study participation.

The endoscopists assigned to the intervention arm will be invited to take part in one training session designed in Phase I of the study (according to the evaluation questionnaire from Phase I). Willing overperformers will be asked to participate in the training as teachers. The training session will be divided into two parts: theoretical - presentation of research on painless colonoscopy - and practical - colonoscopy performance with commentary. Subjects matched 1:1 with trainers will take part in such a session, supervised by the study coordinator.

Each endoscopist who underwent training in the second phase of the study will be sent a written, customized feedback on changes after the intervention and information about factors to improve (as per evaluation questionnaire from Phase I of the study). All endoscopists enrolled into Phase II will be followed through PCSP database for the endpoint of painful colonoscopy rate; the intervention arm will be compared with the control group at 6 and 12 months after feedback in order to investigate whether the adjusted painful colonoscopy rate improved as a result of the intervention.

DETAILED DESCRIPTION:
Background and study rationale:

Colorectal cancer (CRC) is the second leading cause of death from cancer in Europe. Several modalities of CRC screening exist, with each screening modality including colonoscopy either as a primary or secondary test (following positive sigmoidoscopy or faecal occult blood test). Unfortunately, patients perceive colonoscopy as a painful and unpleasant procedure. This is one of the major barriers for participation in CRC screening, particularly since those being screened are usually healthy and asymptomatic. Monitoring patient-reported outcomes is one of the understudied performance measures for quality in colonoscopy according to recent guidelines.

Since 2014, the Polish Colorectal Cancer Screening Programme (PCSP) has routinely used the Gastronet questionnaire to measure patient-reported outcomes. The Gastronet is a Norwegian quality-assurance programme that was initiated in 2003. Patients fill in the questionnaire at home 1 day after colonoscopy and send it back via traditional mail. Questions on pain are answered on a 4-point scale: no pain, slight pain, moderate pain, and severe pain. This scale has been validated previously.

In previous analysis, the investigators have identified several, independent risk factors for painful colonoscopy. However, the single, most important risk factor for painful colonoscopy was the endoscopist himself. This was shown with regards to pain rates adjusted for all factors found relevant in multivariate models (including sedation). The variation among endoscopists was observed as 11- to 23-fold difference in adjusted painful colonoscopy rate. Adjusting for most measurable variables allowed us to cancel the effect of patient selection or other technical issues (endoscope used etc.) and attribute the observed differences, with high probability, to the individual, unquantifiable technical and nontechnical skills possessed by each endoscopist. These skills comprise both the interpersonal skills required to establish a meaningful patient-endoscopist relationship and individual manual skills.

Among modifiable factors, propofol sedation resulted in better procedure tolerance. In most countries, the propofol sedation must be performed by an anaesthesiologist. This practice generates higher costs and reduces colonoscopy unit capacity, as it requires more time, resources, and personnel. Moreover, sedated colonoscopy poses a greater risk of sedation-related (e.g., pneumonia and cardiovascular events) and procedure-related (e.g., bowel perforation and bleeding) complications. What was surprising, sedation based on combination of opioids and benzodiazepines (regarded devoid of aforementioned downsides of propofol sedation) did not improve colonoscopy tolerance in comparison to no sedation at all. This observation led us to suggesting that only propofol sedation should be regarded as effective in case of colonoscopy.

Taking into account the fact that propofol sedation is not a universal and ultimate remedy to increase colonoscopy satisfaction, directed training should be considered to reduce the rate of painful colonoscopies. Technical and nontechnical skills can be either improved or developed with such training, which should focus not only on reducing the odds for pain during, but also after colonoscopy. Such training is necessary especially in cases of countries with limited colonoscopy and/or anaesthesia services capacity.

Up to date, there are no studies assessing the efficacy of training, aiming at reducing the odds of painful colonoscopy. Moreover, there is no existing data on how such training should be designed. Therefore the investigators propose a two-step study:

1. to design a dedicated training program and
2. to evaluate effectiveness of such training in a randomized controlled trial.

Hypothesis:

Dedicated training reduces the painful colonoscopy rate.

Aim:

To investigate, whether directed training leads to reduction in painful colonoscopy rate.

Methods:

The study will be conducted in two phases:

I. Endoscopist categorization based on their performance with regards to colonoscopy pain (under- over- and average performers), according to feedback provided for colonoscopies before study entry and design of training II. Randomized controlled trial evaluating training effectiveness. Phase I - training (intervention) design The first phase of the study consists of the endoscopist categorization, observation of work and workshop with selected PCSP endoscopists to design the training program.

First of all, to categorize endoscopists, the investigators will build multivariate models (as in our previous work) for dataset from years 2014-2018 for pain during endoscopy, allowing us to divide endoscopists into three categories:

1. Underperformers: endoscopists performing worse than expected (with adjusted painful colonoscopy rate higher than mean).
2. Overperformers: endoscopists performing better than expected (with adjusted painful colonoscopy rate lower than mean).
3. Average performers: endoscopists performing inside the confidence interval for mean adjusted painful colonoscopy rate.

For the purpose of creating dedicated assessment questionnaire, the investigators will adapt existing DOPS questionnaire, with tailored modifications (utilising such categories as loop formation and loop reduction, going through flexures, time to caecum, utilisation of additional techniques (change of position, assistance), non-technical skills (communicating with a patient), time slot for colonoscopy, equipment, assistant involvement, sedation etc.) based on experts' opinions, working in PCSP coordinating centre. First, each expert endoscopist will be asked to suggest 5 key, specific elements that are crucial for painless colonoscopy. These elements will be compiled into one list and divided into appropriate domains (pre-procedure, technical considerations, non-technical skills, infrastructure, etc.). The elements will be formatted into questions with binary answer (yes/no). Next, the investigators will perform visits at willing sites, where screening colonoscopies are done by up to 5 under- or overperformers. During such visits, endoscopists will be assessed during their routine work, in friendly environment, utilising the questionnaire, however the purpose of the visits is to modify the questionnaire, to include aspects not initially covered.

Phase II - randomized controlled trial The second phase of the study consists of the randomized controlled trial evaluating the effectiveness of the training developed in Phase I, based on constructed questionnaire. Endoscopists previously categorized as underperformers and average performers from PCSP screening centres will be randomized in 1:1 ratio either to control arm (practice as usual) or training intervention arm. Overperformers will be asked to participate in training sessions as regular participants, however overperformers will not be randomized and treated as study subjects; after intervention, they will be informed about the study design and training session purpose. The endoscopists assigned to the training intervention group will be invited to take part in one training session, similar to the one introduced in Train Colonoscopy Leaders trial (evaluation questionnaire from Phase I will be used). After the training session, each endoscopist from the intervention arm will be sent a written report, including customized feedback on performance and suggested areas of improvement (on the basis of evaluation questionnaire from Phase I of the study). Endoscopists from the intervention group will be followed through PCSP database and will be compared with the control group at 6 and 12 months after feedback. Endoscopists from the control group will not be trained nor will they be informed about study participation. They will receive a reminder, that dedicated report on painful colonoscopy rate is provided in the PCSP database and they will be monitored for endpoints through PCSP database.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists contributing to Polish Colonoscopy Screening Program
* Endoscopists classified as underperformers and average performers, i.e. endoscopists performing above the adjusted mean rate of painful colonoscopies (with high adjusted painful colonoscopy rate), outside of confidence interval of 99% based on the number of performed colonoscopies, and performing inside the confidence interval of 99%, respectively.
* Colonoscopy volume of at least 100 colonoscopies/year for at least 2 years prior to the study inclusion

Exclusion Criteria:

* Endoscopists from the PCSP coordinating centre
* Endoscopists who have participated in the first phase of the study
* Endoscopists classified as overperformers, i.e. performing below the adjusted mean rate of painful colonoscopies (with high adjusted painful colonoscopy rate), outside of confidence interval of 99% based on the number of performed colonoscopies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Endoscopist adjusted painful colonoscopy rate change | assessed 6 and 12 months after training intervention
  Endoscopist adjusted painful colonoscopy rate change (pain during colonoscopy) assessed 6 and 12 months after training intervention.

SECONDARY OUTCOMES:
Endoscopist adjusted painful colonoscopy rate change - pain after colonoscopy | assessed 6 and 12 months after training intervention
  Endoscopist adjusted painful colonoscopy rate change (pain after colonoscopy) assessed 6 and 12 months after training intervention.
Adenoma detection rate (ADR) | assessed 6 and 12 months after training intervention
  Adenoma detection rate - percentage of colonoscopies with at least one adenoma identified.
Cecum intubation rate (CIR) | assessed 6 and 12 months after training intervention
  Percentage of colonoscopies with cecum reached.
Adjusted painful colonoscopy rate for screening centres (in which assessed endoscopists are working) | assessed 6 and 12 months after training intervention
  Center adjusted painful colonoscopy rate change (pain during colonoscopy) assessed 6 and 12 months after training intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaminski MF, Anderson J, Valori R, Kraszewska E, Rupinski M, Pachlewski J, Wronska E, Bretthauer M, Thomas-Gibson S, Kuipers EJ, Regula J. Leadership training to improve adenoma detection rate in screening colonoscopy: a randomised trial. Gut. 2016 Apr;65(4):616-24. doi: 10.1136/gutjnl-2014-307503. Epub 2015 Feb 10. PMID 25670810